CLINICAL TRIAL: NCT05253573
Title: Mobile Health Technology for Personalized Tobacco Cessation Support Among Cancer Survivors in Laos
Acronym: SurvLaos
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Oklahoma (Other)
Collaborators: Setthathirath Hospital (Other); Lao National Cancer Center (Other); National Center for Laboratory and Epidemiology, Lao PDR (Other); National Tobacco Control Committee, Lao PDR (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB 14125; 3R21CA253600-02S1 (NIH)
Record Dates: First submitted 2022-01-18; First posted 2022-02-24 (Actual); Results first posted 2024-08-28 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Cigarette Smoking
MeSH Terms: conditions — Cigarette Smoking | interventions — Tobacco Use Cessation Devices

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Automated Treatment (Experimental): AT consists of all SC components plus a fully automated smartphone-based JITAI that involves proactive, interactive, and personalized messages, images, or videos in Lao.
  Interventions: Drug: Nicotine patch; Behavioral: Self-help materials (to support smoking cessation); Behavioral: Smartphone-based automated treatment for smoking cessation
- Standard Care (Active Comparator): SC consists of brief advice to quit smoking delivered by research staff, self-help written materials (the WHO's "A guide for tobacco users to quit" that we have translated to and validated in Lao), and a 2-week supply of NRT (transdermal patches).
  Interventions: Drug: Nicotine patch; Behavioral: Self-help materials (to support smoking cessation)

INTERVENTIONS:
Drug: Nicotine patch — Provision of nicotine replacement medications in the form of transdermal patches is important to address nicotine withdrawal/craving for smokers who want to quit. Evidence supporting the safety and efficacy of NRT is vast. The PHS Guideline indicates that use of NRT doubles quit rates and should be considered the minimal standard care. Therefore, we will provide NRT to all participants in both groups in the early cessation phase.
Behavioral: Self-help materials (to support smoking cessation) — Our team has translated and validated the World Health Organization's "A guide for tobacco users to quit" into Lao language for use as the self-help material in this study.
Behavioral: Smartphone-based automated treatment for smoking cessation — The automated treatment(AT) include text messages, images, and videos. The AT content is designed to tap the theoretical mechanisms described in the Phase-Based Model (PBM). That is, treatment content is designed to increase motivation, self-efficacy, use of coping skills, and social support, while reducing nicotine withdrawal symptoms and stress. The AT will begin immediately after enrollment and continue for a 12-week period. The AT approach allows for several levels of personalization for each participant, including tailoring to participants' specific health conditions, individual cessation phases, and participants' self-efficacy level or smoking status in the past week.
  Arms: Automated Treatment

SUMMARY:
The parent project (1R21CA253600-01, R21 phase: 9/1/2020-8/31/2022, R33 phase: 9/1/2022-8/31/2025) aims to adapt and evaluate the efficacy of our theoretically and empirically based mobile health (mHealth) technology to help general patients in Lao People's Democratic Republic (Lao PDR) quit smoking cigarettes. This mHealth automated treatment (AT) approach includes a fully automated, interactive, personalized, smartphone-based intervention for behavioral treatment, delivered through our Insight platform.

The purpose of this projects to expand our mHealth-based intervention to address the pressing need for smoking cessation among cancer survivors and their caregivers in Lao PDR. In this project, the investigators will further adapt the AT intervention to ensure that its content is comprehensible and relevant to the target populations (i.e., cancer survivors and caregivers). Then, the investigators will conduct a pilot randomized controlled trial (RCT, N=80) to evaluate the preliminary efficacy of the intervention. Cancer survivors and caregivers of both sexes who smoke will be identified via medical records at the Setthathirath Hospital (SH) and Lao National Cancer Center (LNCC) and recruited. Similar to the parent project's design, participants will be randomized to 1 of 2 treatment groups: standard care (SC) or AT. SC consists of brief advice to quit smoking delivered by research staff, self-help written materials, and a 2-week supply of nicotine patches. AT consists of all SC components plus our fully-automated interactive smartphone-based treatment program, personalized and tailored to cancer survivors or caregivers. The primary RCT outcome is biochemically confirmed self-reported 7-day point prevalence abstinence at 3 months post-study enrollment. The specific aims are as follows:

Aim 1: Evaluate the feasibility of AT in cancer survivors and caregivers. Hypothesis (H1): ≥75% of AT content will be viewed/opened as indicated by digital date/time stamp in Insight.

Aim 2: Evaluate the preliminary efficacy of AT in each cancer survivor/caregiver subgroup. Hypothesis (H2): At the 12-week follow-up, 7-day point prevalence abstinence will be higher in the AT (vs. SC) group.

DETAILED DESCRIPTION:
Stage 1: Further adapt the AT intervention Before conducting the RCT, the investigators will use a multi-step process to adapt our already developed AT intervention for use by the target populations (i.e., cancer survivors and caregivers). These iterative steps include modifying content, user testing and eliciting feedback, and refining. Specifically, the investigators will review all communication messages in the current AT program and modify them to ensure that they are applicable to cancer survivors and caregivers and to both sexes. Then, the investigators will evaluate the AT content applicability, comprehensibility, and linguistic simplicity and clarity with ~10 cancer survivors or caregivers. The investigators will ensure that approximately half of these testing users are women and that the whole testing sample is demographically diverse. Using input and feedback from these testing users, the investigators will revise the AT further if needed. These series of tests and user-feedback sessions to refine the content further and to debug the system will go through an iterative process as needed. AT content taps on theoretical constructs of the Phase-Based Model (PBM)-a theoretical framework specific to smoking cessation used in our JITAI.

Stage 2: The pilot RCT Participant recruitment. Research staff will review medical records of cancer patients receiving care at the 2 hospitals in the past 2 years, screen for their smoking status documented in the records, and contact those who smoked for further screening. To recruit caregivers, research staff will contact random cancer patients who did not smoke and ask if they have a caregiver and if the caregiver smokes. Given the pilot nature of this study, the investigators propose to recruit independent groups of cancer survivors and caregivers who smoke, i.e., no dyads of smokers, to avoid potential interpersonal interactions.

Baseline assessment. Enrolled participants will complete a 45-minute baseline self- or assisted interview, managed and delivered by REDCap. Participants will be randomly assigned to SC or AT by the REDCap randomization module (simple, 1:1). Smartphones will be loaned to participants as needed. All participants will complete a brief training session on smartphone use and the Insight app. The Insight app also includes a help button for instructions on how to use each feature, which participants can review at any time.

Treatment groups. SC consists of brief advice to quit smoking delivered by research staff, self-help written materials (the WHO's "A guide for tobacco users to quit" that the investigators have translated to and validated in Lao), and a 2-week supply of NRT (transdermal patches). AT consists of all SC components plus a fully automated smartphone-based JITAI that involves proactive, interactive, and personalized messages, images, or videos in Lao. Adapted from the parent study and based on the PBM, AT content is designed to increase motivation, self-efficacy, and use of coping skills and reduce nicotine withdrawal symptoms and stress. AT will begin immediately after enrollment and continue for 12 weeks (about 2 messages/images/videos per day, delivered at participants' preferred time). Quit date is set at day 14 post-enrollment for AT and SC participants. JITAI content for AT participants each week will be personalized and tailored to each participant's baseline information (e.g., sex, cancer types, caregiver status, and current health conditions), current PBM phase, and responses to the brief weekly EMAs that drive AT (see Measures). Our AT only targets cigarette smoking because it is the most common type of tobacco used by Lao smokers (95%).

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥18 years
* Self-reported current combustible cigarette smokers (smoked at least 100 cigarettes in lifetime and currently smoke ≥1 cigarette/day)
* Willing to set a quit date within 2 weeks of study enrollment
* Able to provide written informed consent to participate
* Able to read Lao (score ≥4 points on the Rapid Estimate of Adult Literacy in Medicine-Short Form).

Exclusion Criteria:

* History of a medical condition that precludes use of NRT
* Ineligibility to participate based on medical or psychiatric conditions diagnosed by a physician/clinician
* Enrollment in another cessation program or current use of other cessation medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2022-04-20 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thanh C Bui, Principal Investigator — Stephenson Cancer Center, University of Oklahoma Health Sciences Center (OUHSC)
Locations (2):
- Laos (2):
  - Lao National Cancer Center, Vientiane
  - Setthathirath Hospital, Vientiane

IPD SHARING:
Plan to Share IPD: Yes
Deidentified IPD will be shared upon request, with an established data sharing and using agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: After RCT data collection is complete.
Access Criteria: The PI and OUHSC will review data sharing requests. An inter-institutional data sharing and using agreement will be established. Then, deidentified data will be shared via an institutionally-approved secure mechanism.

REFERENCES:
- [Derived] Keopaseuth P, Xangsayarath P, Kulkarni S, Phandouangsy K, Soulaphy C, Alounlungsy P, Dittaphong V, Xayavong D, Vongdala C, Siengsounthone L, Businelle M, Frank-Pearce SG, Vidrine DJ, Vidrine JI, Bui TC. Mobile Health Technology for Personalized Tobacco Cessation Support Among Cancer Survivors and Caregivers in Laos (Project SurvLaos): Protocol for a Pilot Randomized Controlled Trial. JMIR Res Protoc. 2025 Jul 30;14:e66517. doi: 10.2196/66517. PMID 40736921

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total number of 80 participants, cancer survivors and independent caregivers, who smoke were recruited and randomized to treatment. All enrolled caregivers were independent from enrolled cancer patients/survivors (i.e.. no dyads). Therefore, each enrolled participant was unique.
Groups:
- Automated Treatment (AT): AT consists of all SC components plus a fully automated smartphone-based JITAI that involves proactive, interactive, and personalized messages, images, or videos in Lao.
  Nicotine patch: The provision of nicotine replacement medications in the form of transdermal patches is important to address nicotine withdrawal/craving for smokers who want to quit. The PHS Guideline indicates that use of NRT doubles quit rates and should be considered the minimal standard care.
  Self-help materials (to support smoking cessation): Our team has translated and validated the World Health Organization's "A Guide for Tobacco Users to Quit" into Lao language for use as the self-help material in this study.
  Smartphone-based automated treatment for smoking cessation: Automated treatment(AT) includes text messages, images, and videos. The AT content is designed to tap the theoretical mechanisms described in the Phase-Based Model (PBM). That is, treatment content is designed to increase motivation, self-efficacy, use of coping skills, and social support, while reducing nicotine withdrawal symptoms and stress. The AT will begin immediately after enrollment and continue for 12 weeks. The AT approach allows for several levels of personalization for each participant, including tailoring to participants' specific health conditions, individual cessation phases, and participants' self-efficacy level or smoking status in the past week.
Period: Overall Study
Arm/Group | Automated Treatment (AT) | Standard Care
Started | 40 | 40
Cancer Patients/Survivors | 15 | 15
Caregivers | 25 | 25
Completed Cancer Patients/Survivors | 14 | 15
Completed Caregivers | 25 | 25
Completed | 39 | 40
Not Completed | 1 | 0
Not completed — Death | 1 | 0

BASELINE CHARACTERISTICS:
Population: This analysis excludes one participant who died due to their cancer condition.
Groups:
- Automated Treatment: AT consists of all SC components plus a fully automated smartphone-based JITAI that involves proactive, interactive, and personalized messages, images, or videos in Lao.
  Nicotine patch: Provision of nicotine replacement medications in the form of transdermal patches is important to address nicotine withdrawal/craving for smokers who want to quit. The PHS Guideline indicates that use of NRT doubles quit rates and should be considered the minimal standard care. we will provide NRT to all participants in both groups in the early cessation phase.
  Self-help materials: Our team has translated and validated the World Health Organization's "A guide for tobacco users to quit" into Lao language for use as the self-help material in this study.
  Smartphone-based automated treatment for smoking cessation: automated treatment(AT) includes text messages, images, and videos. The AT content is designed to tap the theoretical mechanisms described in the Phase-Based Model. That is, treatment content is designed to increase motivation, self-efficacy, use of coping skills, and social support, while reducing nicotine withdrawal symptoms and stress. AT will begin immediately after enrollment and continue for 12 weeks. The AT approach allows for several levels of personalization for each participant, including tailoring to participants' specific health conditions, individual cessation phases, and participants' self-efficacy level or smoking status in the past week.
- Total: Total of all reporting groups
Arm/Group | Automated Treatment | Standard Care | Total
Number analyzed (Participants) | 39 | 40 | 79
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.74 (12.94) | 45.47 (9.71) | 44.62 (11.38)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  According to Group: Cancer Patients/Survivor Participants - Female | 2 | 1 | 3
  According to Group: Caregiver Participants - Female | 3 | 1 | 4
  According to Group: Cancer Patients/Survivor Participants - Male | 12 | 14 | 26
  According to Group: Caregiver Participants - Male | 22 | 24 | 46
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 2 | 7
  Male | 34 | 38 | 72
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 39 | 40 | 79
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Laos: Urban | 36 | 37 | 73
  Laos: Non-Urban/Town | 3 | 3 | 6
Ethnicity (Asia) [Count of Participants; unit: Participants]
  Lao | 38 | 40 | 78
  Khmou | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Biochemically Verified 7-day Point Prevalence Abstinence at 3 Months
Description: The primary outcome was smoking status at 3 months post-enrollment. Abstinence was defined as biochemically confirmed self-reported 7-day point prevalence abstinence with expired CO <6 ppm. The percentage of participants in each treatment group achieving biochemically verified 7-day point prevalence abstinence at 3 months is reported.
Time Frame: 3 months post enrollment (window for the 3-month follow-up assessment: weeks 10-14).
Measure: Count of Participants; unit: Participants
Groups:
- Automated Treatment: AT consists of all SC components plus a fully automated smartphone-based JITAI that involves proactive, interactive, and personalized messages, images, or videos in Lao.
  Nicotine patch: Provision of nicotine replacement medications in the form of transdermal patches is important to address nicotine withdrawal/craving for smokers who want to quit. The PHS Guideline indicates that use of NRT doubles quit rates and should be considered the minimal standard care. Therefore, we will provide NRT to all participants in both groups in the early cessation phase.
  Self-help materials: Our team has translated and validated the World Health Organization's "A Guide for Tobacco Users to Quit" into Lao language for use as the self-help material in this study.
  Smartphone-based automated treatment for smoking cessation: The automated treatment (AT) includes text messages, images, and videos. The AT content is designed to tap the theoretical mechanisms described in the Phase-Based Model (PBM). That is, treatment content is designed to increase motivation, self-efficacy, use of coping skills, and social support, while reducing nicotine withdrawal symptoms and stress. The AT will begin immediately after enrollment and continue for 12 weeks. The AT approach allows for several levels of personalization for each participant, including tailoring to participants' specific health conditions, individual cessation phases, and participants' self-efficacy level or smoking status in the past week.
Arm/Group | Automated Treatment | Standard Care
Number analyzed (Participants) | 39 | 40
Participants
  Smoking at 3 Months | 10 | 24
  Abstinent at 3 Months | 29 | 16
Statistical Analysis 1: Comparison: Automated Treatment vs Standard Care; The overall number of participants analyzed reflects the cancer survivors and/or independent caregivers. Participants are not represented separately (as cancer survivors or caregivers) for each Arm. This is because the originally proposed statistical data analysis plan did not aim to analyze the data by each group of caregivers versus cancer patients/survivors (because the statistical power would be very low for doing so; Test type: Superiority; Risk Ratio (RR) = 1.85, 95% CI 2-sided [1.21 to 2.83]

2. Primary Outcome: Percentage of Participants Achieving Biochemically Verified 7-day Point Prevalence Abstinence at 3 Months in Each Cancer Survivor/Caregiver Subgroup.
Description: The primary outcome was smoking status at 3 months post-enrollment. Abstinence was defined as biochemically confirmed self-reported 7-day point prevalence abstinence with expired CO <6 ppm. The percentage of cancer survivor/caregiver participants in each treatment group, achieving biochemically verified 7-day point prevalence abstinence at 3 months is reported.
Time Frame: 3 months post-enrollment (window for the 3-month follow-up assessment: weeks 10-14)
Measure: Count of Participants; unit: Participants
Groups:
- Automated Treatment (AT) - Cancer Survivor Participants; Automated Treatment (AT) - Caregiver Participants: AT consists of all SC components plus a fully automated smartphone-based JITAI that involves proactive, interactive, and personalized messages, images, or videos in Lao.
  Nicotine patch: The provision of nicotine replacement medications in the form of transdermal patches is important to address nicotine withdrawal/craving for smokers who want to quit. The PHS Guideline indicates that use of NRT doubles quit rates and should be considered the minimal standard care.
  Self-help materials (to support smoking cessation): Our team has translated and validated the World Health Organization's "A Guide for Tobacco Users to Quit" into Lao language for use as the self-help material in this study.
  Smartphone-based automated treatment for smoking cessation: Automated treatment(AT) includes text messages, images, and videos. The AT content is designed to tap the theoretical mechanisms described in the Phase-Based Model (PBM). That is, treatment content is designed to increase motivation, self-efficacy, use of coping skills, and social support, while reducing nicotine withdrawal symptoms and stress. The AT will begin immediately after enrollment and continue for 12 weeks. The AT approach allows for several levels of personalization for each participant, including tailoring to participants' specific health conditions, individual cessation phases, and participants' self-efficacy level or smoking status in the past week.
- Standard Care - Cancer Survivor Participants; Standard Care - Caregiver Participants: SC consists of brief advice to quit smoking delivered by research staff, self-help written materials (the WHO's "A guide for tobacco users to quit" that we have translated to and validated in Lao), and a 2-week supply of NRT (transdermal patches).
  Nicotine patch: Provision of nicotine replacement medications in the form of transdermal patches is important to address nicotine withdrawal/craving for smokers who want to quit. Evidence supporting the safety and efficacy of NRT is vast. The PHS Guideline indicates that use of NRT doubles quit rates and should be considered the minimal standard care. Therefore, we will provide NRT to all participants in both groups in the early cessation phase.
  Self-help materials (to support smoking cessation): Our team has translated and validated the World Health Organization's "A guide for tobacco users to quit" into Lao language for use as the self-help material in this study.
Arm/Group | Automated Treatment (AT) - Cancer Survivor Participants | Standard Care - Cancer Survivor Participants | Automated Treatment (AT) - Caregiver Participants | Standard Care - Caregiver Participants
Number analyzed (Participants) | 14 | 15 | 25 | 25
Participants
  Smoking at 3 Months | 2 | 5 | 8 | 19
  Abstinent at 3 Months | 12 | 10 | 17 | 6

3. Secondary Outcome: Cigarettes Smoked Per Day at 3-month Follow-up (Quit=0) Among All Participants
Description: At the 3-month follow-up, participants self-reported their average current number of cigarettes smoked per day. For those who quit, the number of cigarettes smoked per day was 0.
Time Frame: In-clinic 3-month follow-up assessments (window: weeks 10-14)
Population: The overall number of participants analyzed in this outcome measure reflects the combined number of cancer survivor and independent caregiver participants.
Measure: Mean (Standard Deviation); unit: Number of cigarettes smoked per day
Arm/Group | Automated Treatment (AT) | Standard Care
Number analyzed (Participants) | 39 | 40
Number of cigarettes smoked per day | 3.64 (6.20) | 6.6 (6.20)

4. Secondary Outcome: Cigarettes Smoked Per Day at 3-month Follow-up Among Participants Who Smoked at 3 Months
Description: At the 3-month follow-up, participants self-reported their average current number of cigarettes smoked per day. This analysis excludes those who quit.
Time Frame: In-clinic 3-month follow-up assessments (window: weeks 10-14)
Measure: Mean (Standard Deviation); unit: Number of cigarettes smoked per day
Arm/Group | Automated Treatment (AT) | Standard Care
Number analyzed (Participants) | 10 | 24
Number of cigarettes smoked per day | 4 (3.60) | 11.05 (5.27)

5. Secondary Outcome: Cigarettes Smoked Per Day at 3-month Follow-up in Each Cancer Survivor/Caregiver Subgroup (Quit=0), Among 'All' Participants
Description: At the 3-month follow-up, participants self-reported their average current number of cigarettes smoked per day. For those who quit, the number of cigarettes smoked per day was 0. This analysis includes all participants in each treatment group.
Time Frame: In-clinic 3-month follow-up assessments (window: weeks 10-14)
Measure: Mean (Standard Deviation); unit: Number of cigarettes smoked per day
Arm/Group | Automated Treatment (AT) - Cancer Survivor Participants | Standard Care - Cancer Survivor Participants | Automated Treatment (AT) - Caregiver Participants | Standard Care - Caregiver Participants
Number analyzed (Participants) | 14 | 15 | 25 | 25
Number of cigarettes smoked per day | 2.85 (5.70) | 2.40 (4.30) | 4.08 (6.53) | 9.12 (5.84)

6. Secondary Outcome: Cigarettes Smoked Per Day at 3-month Follow-up in Each Cancer Survivor/Caregiver Subgroup, Among Participants Who Smoked at 3 Months
Description: At the 3-month follow-up, participants self-reported their average current number of cigarettes smoked per day. This analysis includes only participants in each treatment group who smoked at 3 months. All cancer patients/survivor participants in the Standard Care treatment group self-reported quit smoking at 3 months.
Time Frame: In-clinic 3-month follow-up assessments (window: weeks 10-14)
Population: All cancer patients/survivor participants in the Standard Care treatment group quit smoking at 3 months.
Measure: Mean (Standard Deviation); unit: Number of cigarettes smoked per day
Arm/Group | Automated Treatment (AT) - Cancer Survivor Participants | Standard Care - Cancer Survivor Participants | Automated Treatment (AT) - Caregiver Participants | Standard Care - Caregiver Participants
Number analyzed (Participants) | 1 | 0 | 2 | 19
Number of cigarettes smoked per day | 5 (0) |  | 3.50 (4.94) | 11.05 (5.27)

ADVERSE EVENTS:
Time Frame: 3 months
Description: Adverse event data was collected per arm (Automated treatment and Standard care) and not according to participant groups (caregiver participants and cancer survivor participants). This is because the originally proposed statistical data analysis plan did not aim to analyze the data by each group of caregivers versus cancer patients/survivors (because the statistical power would be very low for doing so).
Arm/Group | Automated Treatment | Standard Care
All-Cause Mortality (participants affected / at risk) | 1/40 | 0/40
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/40
Other Adverse Events (participants affected / at risk) | 0/40 | 0/40

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-03-21): https://cdn.clinicaltrials.gov/large-docs/73/NCT05253573/Prot_SAP_000.pdf